CLINICAL TRIAL: NCT00872378
Title: A Pilot Study of the Effects of BYETTA® (Exenatide) on Weight Loss in Morbidly Obese Non Diabetic Patients Following Adjustable Gastric Banding
Brief Title: The Effects of Exenatide After Gastric Restriction
Acronym: AGREE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Advanced Specialty Care (Other)
Responsible Party: Patrick J. McCarthy M.D., Endocrinologist, Endocrinology Services NorthWest
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASC-AGREE Study
Record Dates: First submitted 2009-03-27; First posted 2009-03-31 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Morbid Obesity
Keywords: Morbid Obesity; LAP Band; Adjustable Gastric Band; Exenatide; Byetta; Weight Loss; Bariatric Surgery
MeSH Terms: conditions — Obesity, Morbid; Weight Loss | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exenatide (Active Comparator): Laparoscopic adjustable gastric banding group: twice daily exenatide therapy plus a standard diet and exercise program
  Interventions: Drug: Exenatide
- Placebo (Placebo Comparator): Laparoscopic adjustable gastric banding group: twice daily placebo therapy plus a standard diet and exercise program
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exenatide — Exenatide titrated up to 20mcg BID. (4 weeks at 5mcg BID; 4 weeks at 10mcg BID; 4 weeks at 15mcg BID; 37 weeks at 20mcg BID).
  Other Names: BYETTA
  Arms: Exenatide
Drug: Placebo — Placebo titrated up to 20mcg BID. (4 weeks at 5mcg BID; 4 weeks at 10mcg BID; 4 weeks at 15mcg BID; 37 weeks at 20mcg BID).
  Arms: Placebo

SUMMARY:
The purpose of this study is to describe change in body weight in non-diabetic morbidly obese patients after laparoscopic adjustable gastric banding (LAGB) with twice daily exenatide or placebo injections.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years,
2. Have a body mass index ≥ 40 kg/m2 or ≥ 35 kg/m2 with comorbidities (1991 NIH Guidelines for Bariatric Surgery),
3. For women of childbearing age, must have a negative pregnancy test at screening, and agree to use barrier contraceptives for the duration of the study, AND
4. Are able to understand and comply with the study process, and give informed consent.

Exclusion Criteria:

1. A diagnosis of type 1 diabetes mellitus,
2. A diagnosis of type 2 diabetes mellitus (A diagnosis of T2DM will be a previous fasting plasma glucose greater than or equal to 126 mg/dL, or a random plasma glucose greater than 200 mg/dL),
3. Have experienced hypersensitivity reaction or a worsening of glycemic control on Byetta® (exenatide),
4. Patients with end stage renal disease or severe renal impairment,
5. Patients with severe gastrointestinal disease, including gastroparesis,
6. Liver function tests 2.5 standard deviations above normal values,
7. Contraindication for bariatric surgery,
8. Treatment with exenatide (Byetta) in the last three months,
9. Currently using or have used within three months before this trial: sibutramine, orlistat, or phentermine(patients must also agree to not use these medications for the duration of the study),
10. Treatment with any investigational drug in the last 30 days,
11. Active malignancy, liver of kidney failure, symptomatic coronary heart disease, or severe psychiatric disease,
12. History of malignancy other than basal cell skin carcinoma, OR
13. In the opinion of the investigator, patient is abusing alcohol and/or drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To describe change in body weight in non-diabetic morbidly obese patients after laparoscopic adjustable gastric banding (LAGB) with twice daily exenatide plus lifestyle modification plan or placebo plus lifestyle modification plan. | 52 weeks

SECONDARY OUTCOMES:
Body Mass Index (BMI) | 52 Weeks
Waist circumference | 52 Weeks
Changes in: 2 hour Oral Glucose Tolerance Test; Lipid panel; Comprehensive metabolic panel; Glycosylated hemoglobin A1c | 52 Weeks
Carotid intima media thickness(CIMT) | 52 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J McCarthy, M.D., Principal Investigator — Endocrinology Services NorthWest
Locations (2):
- United States (2):
  - Advanced Specialty Care, Bend, Oregon
  - Endocrinology Services NorthWest, Bend, Oregon